CLINICAL TRIAL: NCT06822946
Title: Zhibitai Capsules for the Treatment of Primary Hyperlipidemia (Tan yu hu Jie, qi Xue bu li Zheng) A Randomized, Double-blind, Parallel Controlled, Multicenter, Phase II Clinical Trial
Brief Title: Zhibitai Capsules for the Treatment of Primary Hyperlipidemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chengdu Diao Jiuhong Pharmaceutical Factory (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SJTS-20-06-201
Record Dates: First submitted 2025-02-07; First posted 2025-02-12 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Primary Hyperlipidemia
Keywords: zhibitai; primary hyperlipidemia
MeSH Terms: interventions — zhibitai

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental)
  Interventions: Drug: zhibitai capsule
- control group (Active Comparator)
  Interventions: Drug: zhibitai capsule

INTERVENTIONS:
Drug: zhibitai capsule — 2 capsule of Zhibitai capsule/time, 2 times/day, oral
  Arms: Experimental group
Drug: zhibitai capsule — (1 capsule of Zhibitai capsules+1 capsule of Zhibitai capsule simulant)/time, 2 times/day, oral
  Arms: control group

SUMMARY:
Exploring the benefit risk ratio of increase in dosage of Zhibitai capsules (2 capsules at a time, 2 times a day) compared to the original dosage (1 capsule at a time, 1 day)

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 75 years old (inclusive), regardless of gender;
2. BMI (Body Mass Index) between 18.0 kg/m² and 30.0 kg/m²;
3. Meets the diagnostic criteria for primary hyperlipidemia (tan yu hu jie, qi xue bu li zheng);
4. LDL-C level ≥ 3.4 mmol/L and TG level ≤ 4.5 mmol/L;
5. Diagnosis before and after the run-in period meets the above criteria, and the absolute difference between the two LDL-C measurements before and after the run-in period does not exceed 12%;
6. Agrees to follow dietary and lifestyle modification guidance during the trial, maintain a stable diet and exercise routine throughout the study, take medication as required, and complete diary cards;
7. Agrees to participate in this clinical trial and voluntarily signs the informed consent form.

Exclusion Criteria:

1. Known or suspected allergy to any component of the investigational product, or having an allergic constitution.
2. According to the "Chinese Guidelines for Lipid Management (2023)", individuals classified as being at very high risk or extremely high risk for ASCVD.
3. Confirmed homozygous familial hypercholesterolemia.
4. Dyslipidemia caused by secondary reasons, such as nephrotic syndrome, hypothyroidism, renal failure, systemic lupus erythematosus, glycogen storage disease, myeloma, lipodystrophy, acute porphyria, polycystic ovary syndrome, drug-induced causes (e.g., phenothiazines, beta-blockers, glucocorticoids, certain contraceptives, etc.), or patients currently using heparin, thyroid hormone therapy, or other medications that affect lipid metabolism.
5. Any surgical or medical condition that may significantly affect the absorption, distribution, metabolism, or excretion of the drug:

   * History of major gastrointestinal surgery, such as gastrectomy, gastrointestinal anastomosis, or intestinal resection; ② Active or recurrent irritable bowel syndrome (IBS) or inflammatory bowel disease (except for those asymptomatic for at least 6 months prior to the screening visit);

     * Current active gastritis, active ulcer, or gastrointestinal bleeding;

       * History of pancreatic or gallbladder disease (except for those with prior cholecystectomy).
6. Previous use of proprotein convertase subtilisin/kexin type 9 (PCSK9) inhibitors, such as evolocumab and alirocumab.
7. Use of lipid-lowering drugs within 4 weeks prior to enrollment or within 5 half-lives of the drug (whichever is longer), such as statins, cholesterol absorption inhibitors, probucol, bile acid sequestrants, fibrates, niacin, high-purity fish oil preparations, weight-loss drugs (e.g., GLP-1 receptor agonists), and other traditional Chinese medicines, health products, or hospital preparations (e.g., formula granules, herbal decoctions) with clear lipid-lowering effects as stated in the instructions.
8. History of acute or chronic liver disease, drug-induced liver injury, or cirrhosis (except for mild fatty liver indicated by abdominal ultrasound).
9. ALT or AST ≥ 2 times the upper limit of normal (ULN), SCr > ULN, total bilirubin (TBIL) ≥ 1.5 times ULN, creatine kinase ≥ 3 times ULN, or any other laboratory test result (blood routine, urine routine, blood biochemistry) exceeding the ULN, and judged by the investigator as potentially affecting efficacy or safety evaluation.
10. History of any of the following severe cardiovascular or cerebrovascular diseases:

    ① Unstable angina or coronary artery bypass grafting within 3 months prior to the screening visit, or percutaneous coronary intervention.
    * Myocardial infarction, shock, life-threatening arrhythmia, or significant ECG abnormalities (e.g., ST-segment abnormalities, pathological Q waves, abnormal QTc interval, etc.) within 6 months prior to the screening visit.

      * History of left ventricular outflow tract obstruction (e.g., aortic stenosis, idiopathic hypertrophic subaortic stenosis).

        * Heart failure ≥ Class II (NYHA classification) at screening. ⑤ Acute stroke within 6 months prior to the screening visit, excluding asymptomatic stroke.
11. Uncontrolled hypertension (history of hypertension with regular medication, and two consecutive blood pressure measurements ≥ 180/110 mmHg at screening), or history of type 1 diabetes, diabetic ketoacidosis, or uncontrolled type 2 diabetes (HbA1c > 7%).
12. Patients with other severe metabolic diseases.
13. History of myositis, myopathy, or rhabdomyolysis, severe muscle abnormalities, and neuropathy.
14. Thyroid dysfunction (e.g., hyperthyroidism, hypothyroidism, etc.) (except for those judged by the investigator as clinically insignificant).
15. Proven intolerance or inefficacy to HMG-CoA reductase inhibitors.
16. History of malignancy within 5 years prior to the first dose, excluding cervical epithelial carcinoma, squamous cell carcinoma, or basal cell carcinoma of the skin that has been clinically cured for 5 years.
17. Pregnant or lactating women, or individuals of either gender with plans for pregnancy within the next 3 months.
18. Suspected or confirmed history of alcohol, drug, or substance abuse.
19. Individuals with special dietary requirements who cannot adhere to the required diet and exercise control, including but not limited to those following extreme weight-loss diets, undergoing or planning to undergo intense exercise programs (e.g., marathon training, fitness training), or intending to start such training during the trial.
20. Positive for any of the following: hepatitis B virus surface antigen (HBsAg), hepatitis C virus (HCV) antibody, human immunodeficiency virus (HIV) antibody, or syphilis-specific antibody (TPHA).
21. Participation in other interventional clinical trials within the past 3 months.
22. Individuals deemed unsuitable for participation in this clinical trial by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2025-03-27 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
The percentage and absolute changes in serum low-density lipoprotein cholesterol (LDL-C) from baseline after 4, 8, and 12 weeks of treatment | From enrollment to the end of treatment at 4, 8,12 weeks

SECONDARY OUTCOMES:
The proportion of ASCVD low-risk subjects with LDL-C < 3.4 mmol/L after 12 weeks of treatment | From enrollment to the end of treatment at 12 weeks
The proportion of ASCVD medium- and high-risk subjects with LDL-C < 2.6 mmol/L after 12 weeks of treatment | From enrollment to the end of treatment at 12 weeks

OTHER OUTCOMES:
The percentage and absolute changes in total cholesterol (TC) from baseline after 4, 8, and 12 weeks of treatment | From enrollment to the end of treatment at 4,8,12 weeks
The percentage and absolute changes in triglycerides (TG) from baseline after 4, 8, and 12 weeks of treatment | From enrollment to the end of treatment at 4,8,12 weeks
The percentage and absolute changes in high-density lipoprotein cholesterol (HDL-C) and non-HDL-C from baseline after 4, 8, and 12 weeks of treatment | From enrollment to the end of treatment at 4,8,12 weeks
The percentage and absolute changes in Apo A1 and Apo B from baseline after 4, 8, and 12 weeks of treatment | From enrollment to the end of treatment at 4,8,12 weeks
The percentage and absolute changes in lipoprotein(a) [Lp(a)] from baseline after 4, 8, and 12 weeks of treatment | From enrollment to the end of treatment at 4,8,12 weeks
Cure rate, excellent improvement rate, and total effective rate of traditional Chinese medicine syndromes after 4, 8, and 12 weeks of treatment | From enrollment to the end of treatment at 4,8,12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya Second Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No